CLINICAL TRIAL: NCT02382900
Title: Evaluation of a Two-dose Schedule of Quadrivalent Human Papilloma Virus (Types 6, 11, 16, 18) Recombinant Vaccine in 11-year-old Boys in Mexico City (Gardasil® Merck and Co.).
Brief Title: Two-dose Schedule of Quadrivalent HPV Recombinant Vaccine in 11-year-old Boys in Mexico City
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Secretaria de Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Malaquías López Cervantes, Ph D, Universidad Nacional Autonoma de Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 091-2014
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Human Papilloma Virus
Keywords: quadrivalent; vaccine
MeSH Terms: interventions — Vaccines, Synthetic; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): 11 year old boys enrolled in fifth grade of 40 public elementary schools of Mexico City, from the political demarcations of Azcapotzalco, Gustavo A. Madero, Iztacalco, Miguel Hidalgo, Venustiano Carranza, Iztacalco and Tlalpan, reciving a two-dose vaccination scheme (0-6). 250 subjects will be recruited.
  Interventions: Biological: quadrivalent human papillomavirus (types 6, 11, 16,18) recombinant vaccine
- Cohort 2 (Active Comparator): Historical cohort of young women 18-24 years old recruited by Lazcano et. al. receiving a standard vaccination schedule (0-1-6 months). 500 subjects were recruited.
  Interventions: Biological: quadrivalent human papillomavirus (types 6, 11, 16,18) recombinant vaccine
- Cohort 3 (Active Comparator): 11 year old girls enrolled in fifth grade of 40 public elementary schools of Mexico City, from the political demarcations of Azcapotzalco, Venustiano Carranza, Iztacalco and Tlalpan, reciving a two-dose vaccination scheme (0-6). 250 subjects will be recruited.
  Interventions: Biological: quadrivalent human papillomavirus (types 6, 11, 16,18) recombinant vaccine

INTERVENTIONS:
Biological: quadrivalent human papillomavirus (types 6, 11, 16,18) recombinant vaccine — dose scheme (0 and 6 month)
  Other Names: Gardasil

SUMMARY:
In the genital tract human papilloma virus (HPV), especially types 6 and 11 cause genital warts, the commonest viral sexually transmitted disease. The HPV 16 and 18 are the most common oncogenic "high-risk" genotypes and cause approximately 70% of all cervical cancers despite the fact that are associated with other anogenital cancers, anus, vagina, vulva and penis, and cancers of the head and neck. Current estimates are that 5.2% of all cancers are HPV associated. A large number of studies, including both adult and young females, have demonstrated that HPV vaccines are highly immunogenic and induce a long lasting protection against infection. Immunogenic vaccination results in young men and boys are equally satisfactory with the quadrivalent HPV (types 6, 11, 16, 18) vaccine recommended for men. The recommended vaccination scheme includes three shots giving the second at two months and the third at six months after the initial shot. Recently, it has been shown that the use of a two shot scheme (0 and 6 months) is equally effective among girls. The purpose of this study is to determine that the immunogenicity is non-inferior in boys using a two shot scheme compared with young women and girls.

ELIGIBILITY:
Inclusion Criteria:

* All those children whose parents accept their participation in the study.

Exclusion Criteria:

* Fever,
* previous vaccination against HPV,
* allergy to vaccine components,
* thrombocytopenia,
* immunosuppression,
* diarrhea,
* vomiting,
* dyscrasia,
* administration of another anti-viral vaccine in the previous 15 days.

Ages: 10 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity (Geometric mean antibody concentration will be compared between the two groups) | 7 months (1 month after the last dose)
  Geometric means will be compared between the two groups of interest (boys and young women)

CONTACTS AND LOCATIONS:
Locations (1):
- Malaquias Lopez Cervantes, Mexico City, Mexico City, Mexico